CLINICAL TRIAL: NCT04248803
Title: Efficacy of Gluma Desensitizer in Controlling the Immediate Post-treatment Sensitivity in Etch-and-rinse and Self-etch Adhesive Bonded Occlusal Composite Restorations
Brief Title: Evaluation of Gluma Desensitizer in Post-treatment Sensitivity in Posterior Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tamil Nadu Dr.M.G.R.Medical University (Other)
Responsible Party: Principal Investigator, Dr. Geeth Deepika, Principal Investigator, Tamil Nadu Dr.M.G.R.Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSICDSR
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Sensitivity, Tooth
MeSH Terms: conditions — Dentin Sensitivity | interventions — Gluma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Total etch control group (No Intervention): No gluma desensitizer application
- TE - GLUMA application prior to acid etching (Experimental): TE- Total Etch GLUMA - Desensitizing agent
  Interventions: Other: GLUMA (Kulzer GmbH, Germany) desensitizing agent
- TE - GLUMA application after acid etching (Experimental): TE- Total Etch GLUMA - Desensitizing agent
  Interventions: Other: GLUMA (Kulzer GmbH, Germany) desensitizing agent
- Self etch control group (No Intervention): No gluma desensitizer application
- SE - GLUMA application prior to acid etching (Experimental): SE - Self Etch GLUMA - Desensitizing agent
  Interventions: Other: GLUMA (Kulzer GmbH, Germany) desensitizing agent
- SE - GLUMA application after acid etching (Experimental): SE - Self Etch GLUMA - Desensitizing agent
  Interventions: Other: GLUMA (Kulzer GmbH, Germany) desensitizing agent

INTERVENTIONS:
Other: GLUMA (Kulzer GmbH, Germany) desensitizing agent — GLUMA desensitizer is used to reduce tooth sensitivity
  Arms: SE - GLUMA application after acid etching; SE - GLUMA application prior to acid etching; TE - GLUMA application after acid etching; TE - GLUMA application prior to acid etching

SUMMARY:
To evaluate the effect of Gluma desensitizer in controlling immediate post-treatment sensitivity in posterior occlusal composite restorations.

DETAILED DESCRIPTION:
The primary objective of this study is to observe the effect of gluma desensitizer application in controlling the post-treatment sensitivity in posterior occlusal composite restoration in molar teeth using 2 adhesive bonding strategies.

The secondary objective is to evaluate the difference in the post-treatment sensitivity on application of Gluma desensitizer either prior to or after acid etching.

The different adhesive gluma desensitizer application groups are randomly divided into 6 groups,

1. Total etch control group (No gluma desensitizer application)
2. Total etch group Gluma (Kulzer GmbH, Germany) desensitizer application prior to acid etching
3. Total etch group Gluma (Kulzer GmbH, Germany) desensitizer application after acid etching
4. Self etch control group (No gluma desensitizer application)
5. Self etch group Gluma (Kulzer GmbH, Germany) desensitizer application prior to acid etching
6. Self etch group Gluma (Kulzer GmbH, Germany) desensitizer application after acid etching

ELIGIBILITY:
Inclusion Criteria:

* Occlusal cavitated caries in maxillary and mandibular first and second molars

Exclusion Criteria:

* Occlusal caries with axial or proximal extension
* Teeth with periodontal treatment within last three months
* Teeth with cracks
* Teeth to be taken as abutment for prosthesis
* Patients with psychiatric treatment
* Patients in orthodontic treatment or going to need orthodontic treatment
* Patients under dentin hypersensitivity or using desensitizer treatment
* Patients not willing for post treatment follow up
* Patients having any other teeth with pain or sensitivity symptoms
* Caries excavation with pulp exposure and post treatment sensitivity due to occusal interference in restoration

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GEETH DEEPIKA, MDS, Principal Investigator — TN MGR MEDICAL UNIVERSITY
Locations (1):
- CSI College of Dental Sciences and Research, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Out Patient Department of Conservative Dentistry and Endodontics with a chief complaint of decayed tooth during the period from 2020 to 2024. The first patient was enrolled on February 6,2020 and the last patient was enrolled on February 20, 2025
Pre-assignment Details: Of 570 enrolled participants, out of these 546 met the inclusion criteria and were randomized to study groups
Groups:
- Total Etch (TE) Control Group; Self Etch (SE) Control Group: No gluma desensitizer application
Period: Overall Study
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Started | 91 | 91 | 91 | 91 | 91 | 91
Completed | 84 | 84 | 84 | 84 | 84 | 84
Not Completed | 7 | 7 | 7 | 7 | 7 | 7
Not completed — Lost to Follow-up | 7 | 7 | 7 | 7 | 7 | 7

BASELINE CHARACTERISTICS:
Population: A total of 570 participants were enrolled for the study of which only 546 participants met the inclusion criteria which is been described earlier. The participants who met the inclusion criteria were randomly assigned to 6 study groups with 91 participants in each group
Groups:
- Total Etch (TE)Control Group; Self Etch (SE) Control Group: No gluma desensitizer application
- Total: Total of all reporting groups
Arm/Group | Total Etch (TE)Control Group | TE - GLUMA Application Prior to Acid Etching | TE - GLUMA Application After Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching | Total
Number analyzed (Participants) | 91 | 91 | 91 | 91 | 91 | 91 | 546
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8) | 28 (8) | 27 (8) | 28 (9) | 30 (8) | 27 (7) | 28.37 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 39 | 28 | 42 | 10 | 35 | 183
  Male | 62 | 52 | 63 | 49 | 81 | 56 | 363
Race (NIH/OMB) [Count of Participants; unit: Participants] — All participants belong to the Indian Subcontinent (Asian).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 91 | 91 | 91 | 91 | 91 | 91 | 546
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 91 | 91 | 91 | 91 | 91 | 91 | 546
Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — A Visual Analogue Scale (VAS) is one of the pain rating scale ranging from 1 to 10 the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. From the patient's perspective, this spectrum appears continuous. often categorized as none (VAS=0), mild (VAS=1-3), moderate (VAS=4-6)and severe (VAS=7-10). VAS is widely used due to its simplicity and adaptability to a broad range of populations and settings.
  units on a scale | 0.86 (1.67) | 1.72 (2.15) | 1.16 (2.07) | 1.88 (2.25) | 0.63 (1.05) | 2.11 (2.40) | 1.39 (1.93)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Sensitivity Having VAS Score >3
Description: post-operative sensitivity is evaluated using Visual Analog Scale(VAS) VAS rating Score (1 to 10): 1-3: Mild, 4-6:Moderate,7-10:Severe
Time Frame: 24 hours
Population: 84 participants in each group were analyzed for post operative sensitivity using visual analogue scale (VAS) ranging from 1 -10 at the end of 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84
Participants | 14 | 12 | 6 | 16 | 15 | 21
Statistical Analysis 1: Comparison: Total Etch (TE) Control Group vs TE - GLUMA Application After Acid Etching vs TE - GLUMA Application Prior to Acid Etching vs Self Etch (SE) Control Group vs SE - GLUMA Application Prior to Acid Etching vs SE - GLUMA Application After Acid Etching; The sample size was estimated to be 504 using G Power software with 95% power and alpha value set to 0.05. The participants were randomly divided to 6 groups with randomizer.org. The statistical analysis was carried out using SPSS 23 software to compare the mean pain scores between the six study groups using kruskal Wallis test; Test type: Non-Inferiority — From the above mentioned non inferiority clinical trial it is hypothesized that GLUMA application will reduce postoperative sensitivity during dental restorative procedures; p = 0.05, Kruskal-Wallis

2. Primary Outcome: Number of Participants With Post-operative Sensitivity Having VAS Score >3
Description: as for outcome 1
Time Frame: 48 hours
Population: 84 participants in each group were analyzed for post operative sensitivity using VAS ranging from 1 - 10 at the end of 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84
Participants | 14 | 12 | 6 | 13 | 4 | 11

3. Primary Outcome: Number of Participants With Post-operative Sensitivity Having VAS Score >3
Description: post-operative sensitivity is evaluated using Visual Analog Scale(VAS) and cold spray VAS rating Score (1 to 10): 1-3: Mild, 4-6:Moderate,7-10:Severe
Time Frame: 1 week
Population: 84 participants in each group were analyzed for post operative sensitivity using VAS ranging from 1 - 10 at the end of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84
Participants | 6 | 12 | 3 | 9 | 2 | 12

4. Secondary Outcome: Number of Participants With Stimulus Based/ Spontaneous Post-operative Sensitivity Having VAS Score >3
Description: post-operative sensitivity is either due to stimulus or spontaneous is evaluated using Visual Analog Scale(VAS) VAS rating Score (1 to 10): 1-3: Mild, 4-6:Moderate,7-10:Severe
Time Frame: 24 hours
Population: Post operative sensitivity either stimulus based or spontaneous were analyzed using VAS ranging from 1 - 10 at the end of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84
Participants | 14 | 12 | 6 | 16 | 15 | 7

5. Secondary Outcome: Number of Participants With Stimulus Based/ Spontaneous Post-operative Sensitivity Having VAS Score >3
Description: as for outcome 4
Time Frame: 48 hours
Population: Post operative sensitivity either stimulus based or spontaneous were analyzed using VAS ranging from 1 - 10 at the end of 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84
Participants | 14 | 12 | 6 | 13 | 4 | 3

6. Secondary Outcome: Number of Participants With Stimulus Based/ Spontaneous Post-operative Sensitivity Having VAS Score >3
Description: as for outcome 4
Time Frame: 1 week
Population: Post operative sensitivity either stimulus based or spontaneous were analyzed using VAS ranging from 1 - 10 at the end of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Total Etch (TE) Control Group | TE - GLUMA Application After Acid Etching | TE - GLUMA Application Prior to Acid Etching | Self Etch (SE) Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
Number analyzed (Participants) | 84 | 84 | 84 | 84 | 84 | 84
Participants | 6 | 6 | 6 | 7 | 2 | 2

ADVERSE EVENTS:
Time Frame: The study began enrolling participants from February 6, 2020 to February 20, 2025. The adverse events were thoroughly examined for each participant who was enrolled in this clinical trial started from their baseline period at the end of 24 hours till their final visit at the end of 1 week. The last participant was recruited on February 13, 2025 and adverse events were examined with the study completion on February 20, 2025. The adverse events time frame for this study would be "1 Week".
Arm/Group | Total Etch Control Group | TE - GLUMA Application Prior to Acid Etching | TE - GLUMA Application After Acid Etching | Self Etch Control Group | SE - GLUMA Application Prior to Acid Etching | SE - GLUMA Application After Acid Etching
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/84 | 0/84 | 0/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/84 | 0/84 | 0/84 | 0/84
Other Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/84 | 0/84 | 0/84 | 0/84

LIMITATIONS AND CAVEATS:
1. Limited generalizability owing to similar ethnicity and race among all the study participants.
2. Limited reliability of subjective scales such as VAS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs of the current study have no sponsors. (Self-sponsored study)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04248803/Prot_SAP_000.pdf